CLINICAL TRIAL: NCT05163574
Title: Induction of Sustained Unresponsiveness to Peanuts Using High- and Low-dose Peanut Oral Immunotherapy - Evaluation of Efficacy and Safety
Brief Title: Induction of Sustained Unresponsiveness to Peanuts Using High- and Low-dose Peanut Oral Immunotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sustained unresponsiveness
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Peanut Allergy
Keywords: peanut; food allergy; sustained unresponsiveness; children
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose (Experimental): 20 patients
  Interventions: Dietary Supplement: High dose OIT
- Low dose (Active Comparator): 20 patients
  Interventions: Dietary Supplement: Low dose OIT

INTERVENTIONS:
Dietary Supplement: High dose OIT — Patients will receive daily a high dose of peanut flour (300 mg peanut protein) mixed with well-tolerated fruit mousse.
  Arms: High dose
Dietary Supplement: Low dose OIT — Patients will receive daily a low dose of peanut flour (150 mg peanut protein) mixed with well-tolerated fruit mousse.
  Arms: Low dose

SUMMARY:
This study is a continuation of a clinical trial NCT044155930 comparing the efficacy and safety of oral immunotherapy (OIT) with low or high doses of peanut protein (150 or 300 mg, respectively) and will involve patients who have accomplished their per-protocol participation in that trial.

The aim of current study is to assess a sustained unresponsiveness (SU) to allergen protein after at least 8 months of previously assigned high- or low-dose peanut OIT, followed by 4-week-allergen avoidance, and verified by an open oral food challenge (OOFC).

DETAILED DESCRIPTION:
Oral immunotherapy is considered the most effective food allergy treatment. There are two main goals of food immunotherapy: achievement of desensitisation and sustained unresponsiveness. Desensitization is a temporary state of clinical non-reactivity which requires regular intake of allergen, whereas sustained unresponsiveness is defined as lack of clinical reaction to a food allergen after discontinuing OIT for a specific period of time.

The study is a continuation of a clinical trial NCT044155930, which was designed to compare the efficacy and safety of oral immunotherapy (OIT) with low or high doses of peanut protein (150 or 300 mg, respectively) in children with a confirmed diagnosis of peanut allergy. The participants of current study will be recruited from patients who have accomplished their per-protocol participation in previous trial.

Patients will receive the same maintenance dose of peanut allergen, which was used in previous trial (150 or 300 mg, respectively), for at least 8 months (32 weeks +/-2 weeks). Then, OIT will be discontinued for 4 weeks with strict peanut avoidance. After this period, an open oral food challenge (OOFC) will be performed to assess the achievement of sustained unresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* patients who have accomplished their per-protocol participation in trial NCT044155930.
* signed Informed Consent by parent/legal guardian and patient aged>16 years old
* patient's/caregiver's cooperation with researcher

Exclusion Criteria:

* severe asthma
* uncontrolled mild/moderate asthma: forced expiratory volume at one second (FEV1)<80% (under 5 percentile), FEV1/forced vital capacity (FEV)<75% (under 5 percentile), hospitalization due to asthma exacerbation within last 12 months
* current oral/sublingual/subcutaneous immunotherapy with another allergen
* eosinophilic esophagitis
* allergic reaction of 4th or higher grade according to the World Allergy Organisation Systemic Allergic Reaction Grading System during immunotherapy
* a history of severe recurrent anaphylaxis episodes
* chronic diseases requiring continous treatment, including heart disease, epilepsy, metabolic disease, diabetes
* medication:

  * oral, daily steroid therapy exceeding 1 month within the last 12 months
  * at least two courses of oral steroid therapy (at least 7 days) within the last 12 months
  * oral steroid therapy longer than 7 days within the last 3 months
  * biological treatment
  * the need to constantly take antihistamines
  * therapy with b-blockers, angiotensin converting enzyme (ACE) inhibitors, calcium channel inhibitors
* pregnancy
* no consent to participate in the study
* lack of patient cooperation

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Sustained unresponsiveness to a peanut protein after discontinuing oral immunotherapy for 4 weeks. | Up to 9 months after starting maintenance phase
  The share of participants who tolerate a single dose of 150 mg or 300 mg of peanut protein (depending on the maintenance dose) at oral food challenge.
The highest tolerated dose of peanut protein after discontinuing oral immunotherapy for 4 weeks. | Up to 9 months after starting maintenance phase
  Sustained unresponsiveness assessed as the highest tolerated dose of peanut protein at oral food challenge.

SECONDARY OUTCOMES:
Adverse events | Up to 9 months after starting maintenance phase
  Number and severity of adverse events during OIT treatment and at OOFC will be assessed and compared between both groups.
Occurence of eosinophilic esophagitis. | Up to 9 months after starting maintenance phase
  Number and severity of eosinophilic esophagitis symptoms following OIT treatment assessed and compared between both groups.
Laboratory data | Up to 9 months after starting maintenance phase
  Change in serum levels of specific immunoglobulin E (sIgE) to peanut components and peanut-specific immunoglobulin G4 (sIgE4) levels at different time points: at the start and at the end of oral immunotherapy, and after 4 weeks of allergen avoidance, assessed for each individual and compared between groups.
Skin prick test (SPT) | Up to 9 months after starting maintenance phase
  Change in peanut skin prick test wheal in different time points: at the start, and at the end of oral immunotherapy, and after 4 weeks of allergen avoidance, assessed for each individual and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grzela, MD, PhD, Study Chair — Medical University of Warsaw
Locations (1):
- Department of Pediatric Pneumonology and Allergy, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burks AW, Sampson HA, Plaut M, Lack G, Akdis CA. Treatment for food allergy. J Allergy Clin Immunol. 2018 Jan;141(1):1-9. doi: 10.1016/j.jaci.2017.11.004. PMID 29307409
- [Background] Nagakura KI, Yanagida N, Sato S, Nishino M, Asaumi T, Ogura K, Ebisawa M. Low-dose oral immunotherapy for children with anaphylactic peanut allergy in Japan. Pediatr Allergy Immunol. 2018 Aug;29(5):512-518. doi: 10.1111/pai.12898. Epub 2018 May 10. PMID 29603410
- [Background] PALISADE Group of Clinical Investigators; Vickery BP, Vereda A, Casale TB, Beyer K, du Toit G, Hourihane JO, Jones SM, Shreffler WG, Marcantonio A, Zawadzki R, Sher L, Carr WW, Fineman S, Greos L, Rachid R, Ibanez MD, Tilles S, Assa'ad AH, Nilsson C, Rupp N, Welch MJ, Sussman G, Chinthrajah S, Blumchen K, Sher E, Spergel JM, Leickly FE, Zielen S, Wang J, Sanders GM, Wood RA, Cheema A, Bindslev-Jensen C, Leonard S, Kachru R, Johnston DT, Hampel FC Jr, Kim EH, Anagnostou A, Pongracic JA, Ben-Shoshan M, Sharma HP, Stillerman A, Windom HH, Yang WH, Muraro A, Zubeldia JM, Sharma V, Dorsey MJ, Chong HJ, Ohayon J, Bird JA, Carr TF, Siri D, Fernandez-Rivas M, Jeong DK, Fleischer DM, Lieberman JA, Dubois AEJ, Tsoumani M, Ciaccio CE, Portnoy JM, Mansfield LE, Fritz SB, Lanser BJ, Matz J, Oude Elberink HNG, Varshney P, Dilly SG, Adelman DC, Burks AW. AR101 Oral Immunotherapy for Peanut Allergy. N Engl J Med. 2018 Nov 22;379(21):1991-2001. doi: 10.1056/NEJMoa1812856. Epub 2018 Nov 18. PMID 30449234
- [Background] Patrawala M, Shih J, Lee G, Vickery B. Peanut Oral Immunotherapy: a Current Perspective. Curr Allergy Asthma Rep. 2020 Apr 20;20(5):14. doi: 10.1007/s11882-020-00908-6. PMID 32314071
- [Background] Rodriguez Del Rio P, Escudero C, Sanchez-Garcia S, Ibanez MD, Vickery BP. Evaluating primary end points in peanut immunotherapy clinical trials. J Allergy Clin Immunol. 2019 Feb;143(2):494-506. doi: 10.1016/j.jaci.2018.09.035. Epub 2018 Oct 24. PMID 30367908